CLINICAL TRIAL: NCT02097472
Title: A Dose-Finding Study to Assess the Safety, Tolerability, and Immunogenicity of Inactivated Streptococcus Pneumoniae Whole Cell Vaccine Formulated With Alum (PATH-wSP) in Healthy Kenyan Young Adults and PCV-Primed Toddlers
Brief Title: Dose-Finding Study of S.Pneumoniae Whole Cell Vaccine Adsorbed to Alum (PATH-wSP) in Healthy Kenyan Adults and Toddlers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-010
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — PHiD-CV vaccine; 10-valent pneumococcal conjugate vaccine; Pentavac; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Adult Cohort 1, PATH-wSP, 600 mcg (Experimental): A single injection of 600 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 600 mcg PATH-wSP in the alternate arm.
  Interventions: Biological: PATH-wSP
- Adult Cohort 1, Saline (Placebo Comparator): A single injection of saline in one arm, followed 4 weeks later by a single injection of saline in the alternate arm.
  Interventions: Other: Saline
- Adult Cohort 2, PATH-wSP, 1000 mcg (Experimental): A single injection of 1000 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 1000 mcg PATH-wSP in the alternate arm.
  Interventions: Biological: PATH-wSP
- Adult Cohort 2, Saline (Placebo Comparator): A single injection of saline in one arm, followed 4 weeks later by a single injection of saline in the alternate arm.
  Interventions: Other: Saline
- Toddler Cohort 1 PATH-wSP 300 mcg+Active control (Experimental): A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
  Interventions: Biological: PATH-wSP; Biological: Synflorix; Biological: Pentavac
- Toddler Cohort 1 PATH-wSP 300 mcg+Saline (Experimental): A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
  Interventions: Biological: PATH-wSP; Other: Saline
- Toddler Cohort 1: Active Control Only (Active Comparator): A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
  Interventions: Biological: Synflorix; Biological: Pentavac; Other: Saline
- Toddler Cohort 2 PATH-wSP 600 mcg+Active control (Experimental): A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
  Interventions: Biological: PATH-wSP; Biological: Synflorix; Biological: Pentavac
- Toddler Cohort 2 PATH-wSP 600 mcg+saline (Experimental): A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
  Interventions: Biological: PATH-wSP; Other: Saline
- Toddler Cohort 2: Active Control Only (Active Comparator): A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
  Interventions: Biological: Synflorix; Biological: Pentavac; Other: Saline

INTERVENTIONS:
Biological: PATH-wSP — Streptococcus pneumoniae Whole Cell Vaccine adsorbed to Alum
  Arms: Adult Cohort 1, PATH-wSP, 600 mcg; Adult Cohort 2, PATH-wSP, 1000 mcg; Toddler Cohort 1 PATH-wSP 300 mcg+Active control; Toddler Cohort 1 PATH-wSP 300 mcg+Saline; Toddler Cohort 2 PATH-wSP 600 mcg+Active control; Toddler Cohort 2 PATH-wSP 600 mcg+saline
Biological: Synflorix — 1 dose (0.5 mL) contains:
  1 μg of each of the following pneumococcal polysaccharide serotypes:
  1, 5, 6B, 7F, 9V, 14, and 23 F
  And 3 μg of the following pneumococcal polysaccharide serotypes:
  4, 18C and 19F.
  The serotypes are conjugated to either:
  protein D (derived from Non-Typeable Haemophilus influenzae) carrier protein, tetanus toxoid carrier protein or diphtheria toxoid carrier protein
  Other Names: 10-valent Pneumococcal Conjugate Vaccine (PCV10)
  Arms: Toddler Cohort 1 PATH-wSP 300 mcg+Active control; Toddler Cohort 1: Active Control Only; Toddler Cohort 2 PATH-wSP 600 mcg+Active control; Toddler Cohort 2: Active Control Only
Biological: Pentavac — Each PFS contains 0.5 ml (single dose):
  Diphtheria Toxoid 20 Lf to 30 Lf Tetanus Toxoid 2.5 Lf to 10 Lf B. Pertussis 4 IU HBsAg (rDNA) 10 mcg Purified capsular HIB Polysaccharide (PRP) Conjugated to Tetanus Toxoid (carrier protein) 10 mcg Adsorbed on Aluminium Phosphate, AL+++ 1.25 mg Preservative: Thiomersal 0.005 % Dose: O.5ml by intramuscular injection.
  Other Names: Diptheria Pertussis Tetanus Hep B Haemophilus b Conjugate
  Arms: Toddler Cohort 1 PATH-wSP 300 mcg+Active control; Toddler Cohort 1: Active Control Only; Toddler Cohort 2 PATH-wSP 600 mcg+Active control; Toddler Cohort 2: Active Control Only
Other: Saline — 0.9% Sodium Chloride Injection, USP
  Arms: Adult Cohort 1, Saline; Adult Cohort 2, Saline; Toddler Cohort 1 PATH-wSP 300 mcg+Saline; Toddler Cohort 1: Active Control Only; Toddler Cohort 2 PATH-wSP 600 mcg+saline; Toddler Cohort 2: Active Control Only

SUMMARY:
The purpose of this study is to assess the safety and tolerability of PATH-wSP, administered intramuscularly to healthy Kenyan adults and toddlers who have been primed with a pneumococcal conjugate vaccine (PCV).

Additionally, the study will explore whether a measurable immune response is elicited when PATH-wSP is administered to healthy Kenyan adults and toddlers who have been primed with PCV.

DETAILED DESCRIPTION:
S. pneumoniae whole cell vaccine (SPWCV) is a vaccine candidate made from whole, unencapsulated pneumococcal cells. S. pneumoniae whole cell antigen bulk was manufactured at Walter Reed Army Institute of Research from strain RM200 RX1E PdT ΔlytA and is inactivated with beta-propiolactone. Pneumolysin, a proven virulence factor, was genetically knocked out in SPWCV and replaced with pneumolysoid, a derivative carrying the toxin gene with 3 point mutations known to abolish both cytolytic activity and complement activation. When adsorbed to aluminum hydroxide (alum), SPWCV is utilized as the vaccine candidate Streptococcus pneumoniae whole cell vaccine with aluminum hydroxide adjuvant (PATH-wSP) for clinical investigation. PATH-wSP has been previously tested in adults in a Phase 1 trial in the US, in which doses of 100 to 600 μg were given to healthy young adults in a 3-vaccination series and showed a favorable safety, tolerability, and immunogenicity profile.

This study was a dose escalation and age de-escalation study, and sequential cohorts of subjects were identified to allow safety evaluations of dosing and ages to occur progressively during the study. The following PATH-wSP cohorts were defined for adult and toddler subjects:

* Adult Cohort 1: 600 μg PATH-wSP or saline
* Adult Cohort 2: 1000 μg PATH-wSP or saline
* Toddler Cohort 1: 300 μg PATH-wSP and/or active control vaccines
* Toddler Cohort 2: 600 μg PATH-wSP and/or active control vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young Kenyan adults between 18 to 45 years of age
* Willing to provide written informed consent, able to understand comply with study requirements/procedures.
* Adult female subjects surgically sterilized or with a negative serum pregnancy test on enrollment and prior to each vaccination. Adult females must be willing to avoid becoming pregnant over the duration of the study, and must agree to employ an effective form of birth control for the duration of the study.
* Subjects willing to avoid consumption of herbal medication (including herbal medication taken by a mother, which may transmit to a toddler through breast milk) that could have effects on liver function or bleeding indices during the course of the study.
* Healthy toddlers between 12 to 15 months of age who have completed their primary EPI vaccines.
* Toddler's parent willing to provide written informed consent for subject, able to understand and comply with study requirements and procedures.
* Not premature, had a birth weight of >2.5 kg, and a weight-to-height Z score of ≥ -2 at the time of enrollment.

Exclusion Criteria:

* Use of any investigational or nonregistered drug within 90 days prior and during the course of study participation.
* History of administration of any vaccine within 30 days prior to administration of study vaccine or planned vaccination during the course of study.
* History of anaphylactic shock.
* Positive test for malaria (blood film) at time of screening and when retested at Visit 1.
* Immunosuppression or immunodeficiency, inclusive of human immunodeficiency virus, by medical history or by testing at screening.
* Chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or hematological functional abnormality or major congenital defects or illness that requires medical therapy, as deemed by medical history or clinical assessment.
* Evidence of active hepatitis infection (B or C) by immunologic testing at screening.
* Any medical or social condition that in the opinion of the investigator will interfere with the study objectives or pose a risk to the study subject or may prevent the subject from completing the study follow-up.
* An employee (or first degree relative of employee) of the Sponsor, the Clinical Research Organization, or any investigator or site personnel.
* Any screening laboratory test result or vital sign measurement outside normal parameters and deemed by the clinician to be clinically significant, including a positive test for malaria.
* Acute illness (moderate or severe) and/or fever (tympanic temperature >38°C for adults and >37.5°C for toddlers), or any acute and limited illness requiring medical treatment, including the use of antibiotics and treatment for parasites.
* History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines.
* Disorders that require chronic administration of immune-modifying drugs within the past 6 months prior to the administration of the study vaccine.
* Administration of immunoglobulins and/or any blood products within the 6 months preceding enrollment in the study; or anticipation of such administration during the study period.
* Known disturbance of coagulation or other blood disorder in adult subject or in self/first degree relative of toddler subject; or receipt of anticoagulants in the past 3 weeks.
* History of meningitis or seizures or any neurological disorder or major psychiatric disorder (adult).
* Female subjects who are pregnant or breast-feeding.
* Suspicion or recent history of alcohol or substance abuse.
* Toddlers with evidence of congenital abnormality or developmental delay.
* Toddlers with evidence of fetal alcohol syndrome or history of alcohol abuse in mother during pregnancy.
* Toddlers exposed to HIV, born of an HIV infected mother, or who are HIV positive by either antibody or polymerase chain reaction testing.

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nekoye Otsyula, MD, Principal Investigator — Kenya Medical Research Institute/Walter Reed Project
Locations (1):
- Kenya Medical Research Institute/Walter Reed Project, Kisumu, Nyanza, Kenya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: approximately 12 months
  Site: Single center at Kenya Medical Research Institute/Walter Reed Project (KEMRI/WRP) Kombewa Clinical Research Center (CRC)
Groups:
- Adult Cohort 1: PATH-wSP (600 mcg): A single injection of 600 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 600 mcg PATH-wSP in the alternate arm.
- Adult Cohort 2: PATH-wSP (1000 mcg): A single injection of 1000 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 1000 mcg PATH-wSP in the alternate arm.
- Adult Cohort: Saline: A single injection of saline in one arm, followed 4 weeks later by a single injection of saline in the alternate arm.
- Toddler Cohort 1: PATH-wSP (300 mcg)+Active Control: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- Toddler Cohort 1: PATH-wSP (300 mcg)+Saline: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- Toddler Cohort 2: PATH-wSP (600 mcg)+Active Control: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- Toddler Cohort 2: PATH-wSP (600 mcg)+Saline: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- Toddler Cohort: Active Control Only: A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
Period: Received Vaccination 1
Arm/Group | Adult Cohort 1: PATH-wSP (600 mcg) | Adult Cohort 2: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort 1: PATH-wSP (300 mcg)+Active Control | Toddler Cohort 1: PATH-wSP (300 mcg)+Saline | Toddler Cohort 2: PATH-wSP (600 mcg)+Active Control | Toddler Cohort 2: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Started | 18 | 18 | 18 | 50 | 50 | 50 | 50 | 50
Completed | 18 | 18 | 18 | 50 | 50 | 50 | 50 | 50
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Received Vaccination 2
Arm/Group | Adult Cohort 1: PATH-wSP (600 mcg) | Adult Cohort 2: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort 1: PATH-wSP (300 mcg)+Active Control | Toddler Cohort 1: PATH-wSP (300 mcg)+Saline | Toddler Cohort 2: PATH-wSP (600 mcg)+Active Control | Toddler Cohort 2: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Started | 18 | 18 | 18 | 50 | 50 | 50 | 50 | 50
Completed | 18 | 18 | 18 | 50 | 50 | 50 | 49 | 50
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Assessed for Immunogenicity
Arm/Group | Adult Cohort 1: PATH-wSP (600 mcg) | Adult Cohort 2: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort 1: PATH-wSP (300 mcg)+Active Control | Toddler Cohort 1: PATH-wSP (300 mcg)+Saline | Toddler Cohort 2: PATH-wSP (600 mcg)+Active Control | Toddler Cohort 2: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Started | 18 | 18 | 18 | 50 | 50 | 50 | 49 | 50
Completed | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
Not Completed | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adult Cohort: PATH-wSP (600 mcg): A single injection of 600 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 600 mcg PATH-wSP in the alternate arm.
- Adult Cohort: PATH-wSP (1000 mcg): A single injection of 1000 mcg PATH-wSP in one arm, followed 4 weeks later by a single injection of 1000 mcg PATH-wSP in the alternate arm.
- Toddler Cohort: PATH-wSP (300 mcg)+Active Control: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- Toddler Cohort: PATH-wSP (300 mcg)+Saline: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- Toddler Cohort: PATH-wSP (600 mcg)+Active Control: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- Toddler Cohort: PATH-wSP (600 mcg)+Saline: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- Total: Total of all reporting groups
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only | Total
Number analyzed (Participants) | 18 | 18 | 18 | 50 | 50 | 50 | 50 | 50 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.94 (5.98) | 28.56 (8.61) | 30.39 (7.71) | 1.10 (0.09) | 1.09 (0.09) | 1.11 (0.09) | 1.13 (0.10) | 1.09 (0.09) | 5.99 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 7 | 32 | 26 | 23 | 24 | 23 | 148
  Male | 10 | 13 | 11 | 18 | 24 | 27 | 26 | 27 | 156
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 18 | 18 | 18 | 50 | 50 | 50 | 50 | 50 | 304

OUTCOME MEASURES:

1. Primary Outcome: Number/Percent of Adult Subjects Experiencing Fatigue/Malaise Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination.
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Groups:
- PATH-wSP (600 mcg): Vaccination 1: A single injection of 600 mcg PATH-wSP in one arm
- PATH-wSP (1000 mcg): Vaccination 1: A single injection of 1000 mcg PATH-wSP in one arm
- Saline: Vaccination 1: A single injection of saline in one arm.
- PATH-wSP (600 mcg): Vaccination 2: Single injection of 600 mcg PATH-wSP in one arm, one month after initial injection
- PATH-wSP (1000 mcg): Vaccination 2: Single injection of 1000 mcg PATH-wSP in one arm, one month after initial injection
- Saline: Vaccination 2: A single injection of saline in one arm, one month after initial injection
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No fatigue/malaise | 15 | 15 | 18 | 16 | 13 | 15
  Grade 1: no interference with activity | 3 | 3 | 0 | 2 | 2 | 3
  Grade 2: Some interference with activity | 0 | 0 | 0 | 0 | 3 | 0

2. Primary Outcome: Number/Percent of Adult Subjects Experiencing Myalgia Following Vaccination
Description: as for outcome 1
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No myalgia | 11 | 16 | 17 | 15 | 16 | 15
  Grade 1: no interference with activity | 6 | 1 | 1 | 3 | 1 | 3
  Grade 2: Some interference with activity | 1 | 1 | 0 | 0 | 1 | 0

3. Primary Outcome: Number/Percent of Adult Subjects Experiencing Headache Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination.
  Grade 2 includes repeated use of non-narcotic pain reliever for more than 24 hours.
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No headache | 16 | 12 | 13 | 15 | 11 | 12
  Grade 1: no interference with activity | 1 | 6 | 5 | 3 | 6 | 6
  Grade 2: Some interference with activity | 1 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number/Percent of Adult Subjects Experiencing Pain at Injection Site Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination.
  Grade 2 includes use of non-narcotic pain reliever for more than 24 hours.
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No pain at injection site | 4 | 3 | 14 | 9 | 5 | 16
  Grade 1: no interference with activity | 11 | 13 | 4 | 8 | 11 | 2
  Grade 2: Some interference limiting limb use | 3 | 2 | 0 | 1 | 2 | 0

5. Primary Outcome: Number/Percent of Adult Subjects Experiencing Tenderness at Injection Site Following Vaccination
Description: as for outcome 1
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No tenderness | 3 | 4 | 11 | 7 | 7 | 16
  Grade 1: no interference with activity | 12 | 12 | 7 | 10 | 8 | 2
  Grade 2: pain limiting limb use | 3 | 2 | 0 | 1 | 3 | 0

6. Primary Outcome: Number/Percent of Adult Subjects Experiencing Induration at Injection Site Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination.
  Grade 1: does not interfere with activity Grade 2: interferes with activity
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No induration/swelling | 13 | 17 | 17 | 18 | 16 | 18
  Grade 1: 2.5-5cm | 4 | 1 | 1 | 0 | 2 | 0
  Grade 2: 5.1-10cm | 1 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number/Percent of Adult Subjects Experiencing Fever at Injection Site Following Vaccination
Description: as for outcome 1
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 1 | Saline: Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  No fever | 18 | 18 | 18 | 18 | 17 | 18
  Grade 3: ≥39.0 to ≤40.0 degrees Celsius | 0 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Fever Following Vaccination
Description: as for outcome 1
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Groups:
- PATH-wSP (300 mcg)+Active Control: Vaccination 1: A single injection of 300 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh.
- PATH-wSP (300 mcg)+Saline: Vaccination 1: Single injection of 1000 mcg PATH-wSP in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh.
- PATH-wSP (600 mcg)+Active Control: Vaccination 1: A single injection of 600 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh.
- PATH-wSP (600 mcg)+Saline: Vaccination 1: Single injection of 600 mcg PATH-wSP in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh.
- Active Control Only: Vaccination 1: A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh.
- PATH-wSP (300 mcg): Vaccination 2: A single injection of PATH-wSP 300 mcg in the left thigh 8 weeks after the first vaccination of the same dosage
- PATH-wSP (600 mcg): Vaccination 2: A single injection of PATH-wSP 600 mcg in the left thigh 8 weeks after the first vaccination of the same dosage
- Saline: Vaccination 2: A single injection of saline in the left thigh 8 weeks after first vaccination visit of 2 active comparator vaccines (Synflorix and Pentavac) plus 1 saline injection.
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No fever | 26 | 40 | 31 | 42 | 37 | 87 | 78 | 42
  Grade 1: ≥37.5 to ≤38.0 deg. Celsius | 11 | 6 | 13 | 4 | 9 | 5 | 11 | 2
  Grade 2: ≥38.1 to ≤39.0 deg. Celsius | 9 | 3 | 3 | 2 | 3 | 2 | 5 | 2
  Grade 3: ≥39.1 to ≤40.0 deg. Celsius | 3 | 1 | 3 | 2 | 1 | 1 | 0 | 2
  Grade 4: >40.0 deg. Celsius | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Cutaneous Rash Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination.
  Grade 2: includes diffuse macular/maculopapular/morbilliform rash
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No cutaneous rash | 41 | 44 | 43 | 39 | 40 | 83 | 72 | 38
  Grade 1: localized macular rash | 7 | 4 | 5 | 6 | 8 | 9 | 16 | 7
  Grade 2: Diffuse rash or target lesions | 2 | 2 | 2 | 5 | 2 | 3 | 6 | 3

10. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Irritability Following Vaccination
Description: Solicited reactions were assessed for severity during the 60 minutes post vaccination time period, daily for the first week by Field Staff and then at the clinic visit 1 week post vaccination. Severity was defined in the protocol as grade 0-4 (none, mild, moderate, and severe).
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No irritability | 31 | 46 | 36 | 49 | 40 | 90 | 89 | 47
  Grade 1: crying >usual/normal activity | 16 | 4 | 9 | 1 | 9 | 4 | 5 | 1
  Grade 2: crying>usual/interferes w/normal activity | 3 | 0 | 5 | 0 | 1 | 1 | 0 | 0

11. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Drowsiness Following Vaccination
Description: as for outcome 10
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No drowsiness | 48 | 49 | 47 | 50 | 50 | 95 | 94 | 47
  Grade 1: drowsiness easily tolerated | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 2: interferes with normal activity | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

12. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Loss of Appetite Following Vaccination
Description: as for outcome 10
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No loss of appetite | 32 | 42 | 30 | 47 | 31 | 85 | 88 | 45
  Grade 1: eating <usual/normal activity | 17 | 7 | 19 | 3 | 19 | 10 | 6 | 3
  Gr. 2: eating <usual/interferes w/ normal activity | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Pain/Tenderness at Injection Site Following Vaccination
Description: as for outcome 1
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Groups:
- 300 mcg PATH-wSP: Vaccination 1: A single injection of 300 mcg PATH-wSP in the left thigh at first vaccination (during which subjects also received either two saline injections, or or Synflorix and Pentavac injections, in the right thigh)
- 600 mcg PATH-wSP: Vaccination 1: A single injection of 600 mcg PATH-wSP in the left thigh (during which subjects also received either two saline injections, or or Synflorix and Pentavac injections, in the right thigh)
- Active Control: Pentavac: A single injection of the active comparator vaccine Pentavac in the right thigh during the first vaccination.
- Active Control: Synflorix: A single injection of the active comparator vaccine Synflorix in the right thigh during the first vaccination.
- Active Control: Saline: One injection of saline in the left thigh during the first vaccination (during which subjects received Pentavac and Synflorix injections, but no PATH-wSP injections)
- PATH-wSP (300 mcg): Vaccination 2: SA single injection of PATH-wSP 300 mcg in the left thigh 8 weeks after the first vaccination of the same dosage
Arm/Group | 300 mcg PATH-wSP: Vaccination 1 | 600 mcg PATH-wSP: Vaccination 1 | Active Control: Pentavac | Active Control: Synflorix | Active Control: Saline | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 100 | 100 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No pain/tenderness at injection site | 33 | 43 | 17 | 21 | 20 | 72 | 81 | 42
  Grade 1: minor reactions to touch | 61 | 52 | 32 | 28 | 30 | 22 | 13 | 6
  Grade 2: cries/protests to touch | 6 | 5 | 1 | 1 | 0 | 1 | 0 | 0

14. Primary Outcome: Number/Percent of Toddler Subjects Experiencing Induration/Swelling at Injection Site Following Vaccination
Description: as for outcome 10
Time Frame: up to 1 week following first vaccination (Day 7) or second vaccination (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mcg PATH-wSP: Vaccination 1 | 600 mcg PATH-wSP: Vaccination 1 | Active Control: Pentavac | Active Control: Synflorix | Active Control: Saline | PATH-wSP (300 mcg): Vaccination 2 | PATH-wSP (600 mcg): Vaccination 2 | Saline: Vaccination 2
Number analyzed (Participants) | 100 | 100 | 50 | 50 | 50 | 95 | 94 | 48
Participants
  No induration/swelling | 93 | 98 | 45 | 48 | 49 | 93 | 89 | 47
  Grade 1: Induration or edema <2.5cm | 5 | 2 | 4 | 2 | 1 | 2 | 5 | 1
  G2: Induration OR edema ≥2.5cm but <50% surface ar | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against Pneumolysoid (L460D) Pneumococcal Protein: ELISA Assay
Description: Measured with enzyme-linked immunosorbent assay (ELISA).
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 17 | 16 | 46 | 47 | 48 | 47 | 48
titer
  Baseline | 2083.27 [1638.67 to 2648.49] | 1569.91 [1102.09 to 2236.30] | 1998.33 [1356.41 to 2944.02] | 400.00 [289.99 to 551.74] | 311.30 [209.43 to 462.71] | 755.10 [541.85 to 1052.27] | 848.61 [612.56 to 1175.62] | 455.52 [318.02 to 652.45]
  Post-vaccination 1 | 2619.99 [2015.16 to 3406.36] | 2394.59 [1669.66 to 3434.28] | 1945.09 [1329.56 to 2845.58] | 516.79 [367.08 to 727.54] | 506.45 [351.03 to 730.68] | 897.97 [664.86 to 1212.82] | 1647.90 [1208.09 to 2247.81] | 489.62 [355.16 to 674.99]
  Post-vaccination 2 | 3752.62 [2860.91 to 4922.26] | 2933.71 [2049.42 to 4199.55] | 1961.47 [1301.64 to 2955.80] | 800.00 [563.29 to 1136.18] | 732.25 [509.87 to 1051.63] | 1510.20 [1101.94 to 2069.72] | 2211.06 [1592.51 to 3069.87] | 526.28 [386.30 to 716.99]

16. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PspA-Fam1 Pneumococcal Protein: ELISA Assay
Description: Measured with enzyme-linked immunosorbent assay (ELISA).
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 47 | 48
titer
  Baseline | 1899.32 [1393.87 to 2588.06] | 2042.68 [1679.25 to 2484.75] | 1793.44 [1404.90 to 2289.43] | 410.23 [298.75 to 563.30] | 361.41 [268.84 to 485.85] | 550.02 [423.69 to 714.03] | 674.04 [509.70 to 891.36] | 456.64 [349.76 to 596.17]
  Post-vaccination 1 | 2425.50 [1929.04 to 3049.73] | 3083.33 [2532.19 to 3754.44] | 1922.47 [1514.36 to 2440.56] | 565.40 [431.64 to 740.62] | 557.07 [408.19 to 760.24] | 637.63 [495.23 to 820.97] | 1126.67 [831.35 to 1526.90] | 417.09 [309.03 to 562.93]
  Post-vaccination 2 | 3192.07 [2609.98 to 3903.97] | 3901.23 [2943.11 to 5171.26] | 2031.31 [1566.67 to 2633.75] | 724.42 [563.05 to 932.03] | 541.73 [399.29 to 734.98] | 889.48 [707.12 to 1118.86] | 1264.22 [925.59 to 1726.74] | 487.03 [359.40 to 659.99]

17. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against L460D Pneumococcal Protein
Description: Measured using meso scale discovery (MSD).
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: Insufficient sample
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 861.27 [661.13 to 1121.99] | 820.92 [629.25 to 1070.97] | 908.51 [582.64 to 1416.63] | 263.85 [206.73 to 336.74] | 210.15 [160.30 to 275.48] | 309.74 [246.74 to 388.83] | 331.08 [270.14 to 405.77] | 216.45 [173.79 to 269.58]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1127.59 [869.68 to 1461.99] | 998.09 [777.32 to 1281.56] | 886.15 [614.08 to 1278.77] | 329.38 [255.01 to 425.44] | 328.35 [253.48 to 425.33] | 386.92 [316.53 to 472.97] | 602.20 [489.74 to 740.49] | 247.77 [194.90 to 314.98]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1391.66 [1065.65 to 1817.41] | 1410.11 [1014.73 to 1959.55] | 963.25 [701.06 to 1323.49] | 462.54 [351.01 to 609.51] | 408.40 [318.02 to 524.46] | 631.63 [506.72 to 787.32] | 803.61 [630.84 to 1023.69] | 279.43 [221.59 to 352.36]

18. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PspA-Fam1 Pneumococcal Protein: Meso Scale Discovery (MSD) Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 2124.32 [1533.58 to 2942.62] | 2129.61 [1574.00 to 2881.35] | 2049.33 [1457.58 to 2881.30] | 175.80 [122.62 to 252.03] | 174.35 [119.81 to 253.71] | 202.89 [145.92 to 282.09] | 217.24 [154.08 to 306.29] | 177.29 [127.64 to 246.25]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 3149.80 [2268.50 to 4373.47] | 3442.17 [2582.70 to 4587.64] | 2105.22 [1473.42 to 3007.94] | 283.38 [203.73 to 394.15] | 294.98 [203.95 to 426.66] | 272.19 [204.41 to 362.44] | 420.45 [285.84 to 618.44] | 167.21 [112.78 to 247.89]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 3469.35 [2725.55 to 4416.14] | 4607.95 [3491.22 to 6081.90] | 2323.41 [1752.55 to 3080.21] | 367.01 [265.16 to 507.99] | 338.19 [230.39 to 496.43] | 371.56 [279.50 to 493.95] | 518.77 [365.33 to 736.65] | 186.84 [126.04 to 276.97]

19. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PhtD Pneumococcal Protein
Description: Measured using Meso Scale Discovery (MSD) Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 841.63 [626.89 to 1129.94] | 784.56 [606.58 to 1014.75] | 775.26 [531.41 to 1130.99] | 426.11 [313.40 to 579.35] | 403.13 [289.64 to 561.09] | 466.20 [337.37 to 644.21] | 497.28 [383.30 to 645.15] | 434.86 [331.26 to 570.85]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 839.14 [576.12 to 1222.24] | 868.55 [655.40 to 1151.03] | 775.29 [535.14 to 1123.21] | 563.55 [429.28 to 739.83] | 491.70 [361.58 to 668.64] | 577.47 [434.14 to 768.11] | 654.21 [512.33 to 835.39] | 513.83 [390.75 to 675.68]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 890.67 [627.43 to 1264.34] | 982.10 [710.87 to 1356.82] | 872.62 [603.52 to 1261.71] | 804.59 [612.11 to 1057.60] | 704.46 [552.58 to 898.09] | 767.31 [578.07 to 1018.48] | 1074.36 [844.35 to 1367.04] | 679.80 [519.10 to 890.25]

20. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against BCH0785 Pneumococcal Protein
Description: Measured using Meso Scale Discovery (MSD) Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1566.50 [1035.43 to 2369.96] | 1145.05 [909.05 to 1442.33] | 1236.11 [819.09 to 1865.46] | 400.58 [294.10 to 545.61] | 271.66 [200.93 to 367.30] | 281.66 [209.24 to 379.16] | 372.53 [277.67 to 499.79] | 288.13 [206.26 to 402.50]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1665.26 [1070.16 to 2591.29] | 1367.52 [1050.00 to 1781.04] | 1224.22 [787.13 to 1904.02] | 504.49 [372.64 to 682.99] | 364.39 [279.71 to 474.72] | 373.57 [288.65 to 483.48] | 526.34 [385.99 to 717.73] | 328.03 [238.52 to 451.14]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1808.37 [1220.45 to 2679.52] | 1713.83 [1263.06 to 2325.47] | 1340.75 [972.21 to 1849.00] | 561.60 [408.05 to 772.93] | 480.18 [373.03 to 618.11] | 470.01 [350.35 to 630.53] | 716.82 [538.77 to 953.71] | 394.37 [288.87 to 538.41]

21. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against StkP Pneumococcal Protein
Description: Measured using Meso Scale Discovery (MSD) Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1406.04 [901.16 to 2193.77] | 1140.55 [863.69 to 1506.15] | 1263.61 [819.76 to 1947.76] | 204.58 [146.61 to 285.48] | 130.62 [98.14 to 173.85] | 157.58 [113.59 to 218.61] | 229.15 [169.00 to 310.70] | 161.89 [119.32 to 219.65]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1632.87 [1003.67 to 2656.52] | 1311.45 [973.06 to 1767.52] | 1308.29 [825.65 to 2073.06] | 278.64 [204.21 to 380.18] | 164.27 [124.79 to 216.24] | 187.67 [140.60 to 250.51] | 295.14 [219.22 to 397.35] | 180.93 [132.20 to 247.63]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1753.89 [1138.27 to 2702.47] | 1620.05 [1203.93 to 2180.01] | 1430.78 [985.89 to 2076.42] | 351.25 [255.61 to 482.66] | 230.51 [183.42 to 289.68] | 273.84 [205.92 to 364.16] | 396.24 [297.85 to 527.14] | 217.32 [162.69 to 290.28]

22. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PcpA Pneumococcal Protein
Description: Measured using Meso Scale Discovery (MSD) Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1677.20 [1248.67 to 2252.80] | 1016.49 [757.20 to 1364.57] | 1436.97 [996.44 to 2072.26] | 316.39 [202.24 to 494.97] | 350.52 [218.29 to 562.87] | 355.69 [206.59 to 612.41] | 356.24 [224.23 to 565.95] | 254.77 [152.06 to 426.85]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1523.84 [1045.11 to 2221.85] | 904.99 [670.76 to 1221.03] | 1461.34 [1064.83 to 2005.48] | 354.49 [222.21 to 565.50] | 327.75 [203.97 to 526.65] | 473.66 [290.78 to 771.55] | 344.10 [211.00 to 561.19] | 297.33 [181.65 to 486.68]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1497.72 [1127.58 to 1989.36] | 950.83 [668.08 to 1353.25] | 1728.30 [1234.67 to 2419.29] | 375.72 [234.90 to 600.97] | 342.08 [216.65 to 540.12] | 441.77 [265.98 to 733.75] | 434.85 [259.39 to 729.01] | 392.99 [236.60 to 652.75]

23. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against SPWCA Pneumococcal Protein
Description: MSD Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1707.99 [1209.54 to 2411.84] | 1398.09 [969.28 to 2016.60] | 1321.49 [1075.42 to 1623.87] | 664.34 [580.83 to 759.85] | 632.54 [552.55 to 724.12] | 615.81 [530.49 to 714.86] | 665.59 [596.55 to 742.63] | 652.61 [581.79 to 732.04]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1660.20 [1310.34 to 2103.47] | 1359.27 [1049.52 to 1760.45] | 1263.81 [1026.75 to 1555.61] | 778.54 [680.41 to 890.82] | 717.62 [649.35 to 793.07] | 728.65 [639.50 to 830.22] | 771.90 [682.33 to 873.22] | 682.37 [601.34 to 774.32]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1709.46 [1373.92 to 2126.94] | 1685.31 [1318.70 to 2153.85] | 1493.37 [1144.92 to 1947.88] | 844.62 [736.10 to 969.13] | 764.02 [687.93 to 848.52] | 820.14 [739.90 to 909.08] | 939.58 [808.92 to 1091.35] | 765.74 [674.90 to 868.81]

24. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PiuA Pneumococcal Protein
Description: MSD Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1401.11 [895.60 to 2191.93] | 1524.31 [968.09 to 2400.10] | 1625.92 [923.10 to 2863.84] | 677.28 [535.39 to 856.78] | 575.24 [449.63 to 735.94] | 556.30 [442.49 to 699.38] | 679.07 [530.85 to 868.68] | 601.79 [474.76 to 762.80]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 1471.39 [981.61 to 2205.56] | 1668.22 [1077.75 to 2582.20] | 1603.96 [1003.56 to 2563.53] | 837.32 [659.76 to 1062.66] | 732.41 [597.09 to 898.41] | 702.78 [577.60 to 855.08] | 860.69 [672.04 to 1102.30] | 671.40 [526.98 to 855.41]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1582.79 [1021.39 to 2452.74] | 1898.28 [1189.21 to 3030.13] | 1769.43 [1111.95 to 2815.66] | 937.83 [730.15 to 1204.57] | 815.05 [662.34 to 1002.96] | 961.01 [804.64 to 1147.77] | 1108.83 [880.94 to 1395.67] | 763.13 [612.16 to 951.33]

25. Secondary Outcome: Geometric Mean Concentrations (GMC) of IgG Antibodies Against PiaA Pneumococcal Protein
Description: MSD Assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 18 | 18 | 17 | 48 | 50 | 48 | 47 | 49
titer
  Baseline | 1933.77 [1248.16 to 2995.98] | 2027.06 [1481.10 to 2774.27] | 1897.23 [1211.22 to 2971.80] | 650.98 [503.48 to 841.69] | 503.78 [373.57 to 679.38] | 609.28 [476.06 to 779.79] | 892.24 [715.63 to 1112.42] | 542.93 [430.61 to 684.54]
  Post-vaccination 1: number analyzed (Participants) | 18 | 18 | 17 | 48 | 49 | 48 | 47 | 49
  Post-vaccination 1 | 2299.24 [1449.89 to 3646.14] | 2396.09 [1745.84 to 3288.52] | 1853.17 [1231.25 to 2789.21] | 759.91 [605.92 to 953.04] | 622.89 [485.14 to 799.76] | 721.16 [578.45 to 899.08] | 1197.63 [951.41 to 1507.56] | 602.56 [476.30 to 762.28]
  Post-vaccination 2: number analyzed (Participants) | 18 | 17 | 17 | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 2471.44 [1620.81 to 3768.50] | 2875.72 [2003.45 to 4127.76] | 2218.47 [1548.56 to 3178.18] | 926.53 [714.91 to 1200.79] | 833.02 [653.96 to 1061.12] | 880.18 [718.66 to 1078.02] | 1493.50 [1179.45 to 1891.16] | 750.60 [580.03 to 971.33]

26. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against Pneumolysoid (L460D) Pneumococcal Protein: ELISA
Description: Measured using ELISA
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 48
fold change
  Post-vaccination 1 | 1.29 [1.10 to 1.52] | 1.63 [1.34 to 1.98] | 1.19 [1.03 to 1.37] | 1.94 [1.63 to 2.31] | 1.07 [0.89 to 1.29]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 45 | 48
  Post-vaccination 2 | 2.00 [1.60 to 2.49] | 2.35 [1.86 to 2.98] | 2.00 [1.57 to 2.54] | 2.48 [1.88 to 3.28] | 1.16 [0.98 to 1.36]

27. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PspA-Fam1 Pneumococcal Protein: ELISA
Description: Measured using ELISA
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 48
fold change
  Post-vaccination 1 | 1.38 [1.09 to 1.75] | 1.54 [1.28 to 1.85] | 1.16 [0.96 to 1.40] | 1.67 [1.26 to 2.21] | 0.91 [0.79 to 1.06]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.77 [1.39 to 2.24] | 1.50 [1.20 to 1.87] | 1.62 [1.29 to 2.03] | 1.83 [1.34 to 2.49] | 1.07 [0.83 to 1.37]

28. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against Pneumolysoid (L460D) Pneumococcal Protein: MSD
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.25 [1.11 to 1.40] | 1.56 [1.37 to 1.77] | 1.25 [1.14 to 1.37] | 1.82 [1.57 to 2.11] | 1.14 [1.01 to 1.30]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.72 [1.47 to 2.01] | 1.96 [1.66 to 2.31] | 2.04 [1.72 to 2.42] | 2.40 [1.98 to 2.92] | 1.28 [1.11 to 1.48]

29. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PspA-Fam1 Pneumococcal Protein: MSD
Description: Measured using ELISA
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.61 [1.24 to 2.09] | 1.74 [1.48 to 2.04] | 1.34 [1.10 to 1.64] | 1.94 [1.44 to 2.60] | 0.94 [0.80 to 1.11]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 2.09 [1.58 to 2.77] | 1.97 [1.57 to 2.47] | 1.83 [1.46 to 2.29] | 2.38 [1.71 to 3.31] | 1.03 [0.80 to 1.33]

30. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PhtD Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.32 [1.16 to 1.51] | 1.25 [1.11 to 1.42] | 1.24 [0.94 to 1.63] | 1.32 [1.11 to 1.55] | 1.18 [1.04 to 1.34]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.79 [1.53 to 2.09] | 1.90 [1.55 to 2.32] | 1.65 [1.29 to 2.11] | 2.10 [1.73 to 2.56] | 1.60 [1.28 to 1.99]

31. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against BCH0785 Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.26 [1.10 to 1.44] | 1.30 [1.12 to 1.51] | 1.33 [1.08 to 1.63] | 1.41 [1.17 to 1.71] | 1.14 [1.00 to 1.30]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.36 [1.14 to 1.63] | 1.70 [1.41 to 2.05] | 1.67 [1.34 to 2.07] | 1.93 [1.53 to 2.42] | 1.31 [1.05 to 1.64]

32. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against StkP Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.36 [1.19 to 1.56] | 1.26 [1.09 to 1.46] | 1.19 [1.00 to 1.42] | 1.29 [1.12 to 1.48] | 1.12 [1.00 to 1.25]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.69 [1.44 to 1.99] | 1.79 [1.52 to 2.12] | 1.74 [1.40 to 2.15] | 1.67 [1.40 to 2.00] | 1.29 [1.12 to 1.48]

33. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PcpA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.12 [0.91 to 1.39] | 0.95 [0.83 to 1.10] | 1.33 [0.95 to 1.87] | 0.97 [0.73 to 1.28] | 1.17 [0.96 to 1.42]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.17 [0.91 to 1.50] | 1.07 [0.82 to 1.39] | 1.24 [0.92 to 1.68] | 1.17 [0.80 to 1.72] | 1.43 [1.03 to 1.99]

34. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against SPWCA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.17 [1.06 to 1.30] | 1.14 [1.02 to 1.27] | 1.18 [1.05 to 1.34] | 1.16 [1.03 to 1.30] | 1.05 [0.94 to 1.16]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.26 [1.11 to 1.43] | 1.23 [1.10 to 1.38] | 1.33 [1.17 to 1.52] | 1.43 [1.24 to 1.66] | 1.17 [1.04 to 1.31]

35. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PiuA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.24 [1.08 to 1.42] | 1.26 [1.08 to 1.47] | 1.26 [1.05 to 1.52] | 1.27 [1.11 to 1.45] | 1.12 [1.01 to 1.23]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.35 [1.14 to 1.60] | 1.45 [1.23 to 1.74] | 1.73 [1.38 to 2.16] | 1.64 [1.37 to 1.96] | 1.24 [1.07 to 1.42]

36. Secondary Outcome: Geometric Mean Fold Change of IgG Antibodies Against PiaA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: The number analyzed may differ between periods because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
fold change
  Post-vaccination 1 | 1.17 [1.01 to 1.36] | 1.23 [1.03 to 1.47] | 1.18 [1.03 to 1.37] | 1.34 [1.15 to 1.57] | 1.11 [0.98 to 1.26]
  Post-vaccination 2: number analyzed (Participants) | 46 | 47 | 48 | 46 | 48
  Post-vaccination 2 | 1.40 [1.15 to 1.70] | 1.69 [1.32 to 2.16] | 1.44 [1.20 to 1.73] | 1.66 [1.34 to 2.05] | 1.34 [1.11 to 1.62]

37. Secondary Outcome: Fold Change in IgG Response to Pneumolysoid (L460D) Pneumococcal Protein Among Toddler Cohort (ELISA)
Description: Measured using ELISA
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Groups:
- PATH-wSP (300 mcg)+Saline: Vaccination 1: Single injection of 300 mcg PATH-wSP in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh.
- PATH-wSP (300 mcg)+Active Control: Vaccination 2: A single injection of PATH-wSP 300 mcg in the left thigh 8 weeks after the first vaccination of the same dosage plus two active control vaccines in the right thigh.
- PATH-wSP (300 mcg)+Saline: Vaccination 2: Injection of PATH-wSP 300 mcg in the left thigh, 8 weeks after the first vaccination of the same plus a saline injection in the right thigh.
- PATH-wSP (600 mcg)+Active Control: Vaccination 2: A single injection of PATH-wSP 600 mcg in the left thigh, 8 weeks after the first vaccination of the same dosage and two active control vaccinations in the right thigh
- PATH-wSP (600 mcg)+Saline: Vaccination 2: A single injection of 600 mcg PATH-wSP in the left thigh, 8 weeks after receipt of vaccination of the same dosage and two saline injections in the right thigh.
- Active Control Only: Vaccination 2: A single injection of saline in the left thigh, 8 weeks after the same saline injection plus a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh.
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 48 | 46 | 47 | 48 | 45 | 48
Participants
  <2-Fold | 28 | 23 | 32 | 16 | 36 | 18 | 14 | 20 | 14 | 34
  ≥2-Fold | 18 | 24 | 16 | 31 | 12 | 28 | 33 | 28 | 31 | 14

38. Secondary Outcome: Fold Change in IgG Response to PspA-Fam1 (ELISA)
Description: Measured using ELISA
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 48 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 36 | 29 | 42 | 29 | 44 | 30 | 28 | 31 | 25 | 34
  ≥2-Fold | 10 | 18 | 6 | 18 | 4 | 16 | 19 | 17 | 21 | 14

39. Secondary Outcome: Fold Change in IgG Response to L460D Pneumococcal Protein (MSD)
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 48 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 37 | 31 | 43 | 26 | 39 | 23 | 23 | 18 | 6 | 38
  ≥2-Fold, <3-Fold | 8 | 9 | 4 | 13 | 5 | 18 | 14 | 18 | 22 | 8
  ≥3-Fold, <4-Fold | 1 | 4 | 1 | 3 | 2 | 0 | 4 | 3 | 6 | 1
  ≥4-Fold | 0 | 3 | 0 | 5 | 2 | 5 | 6 | 9 | 12 | 1

40. Secondary Outcome: Fold Change in IgG Response to PspA-Fam1 Pneumococcal Protein (MSD)
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 29 | 26 | 35 | 18 | 40 | 16 | 16 | 20 | 4 | 30
  ≥2-Fold, <3-Fold | 12 | 11 | 8 | 15 | 6 | 16 | 21 | 15 | 21 | 11
  ≥3-Fold, <4-Fold | 2 | 7 | 1 | 5 | 2 | 5 | 1 | 4 | 5 | 3
  ≥4-Fold | 5 | 5 | 4 | 9 | 1 | 9 | 9 | 9 | 16 | 4

41. Secondary Outcome: Fold Change in IgG Response to PhtD Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 37 | 39 | 43 | 34 | 42 | 20 | 20 | 22 | 20 | 26
  ≥2-Fold, <3-Fold | 8 | 7 | 3 | 7 | 2 | 18 | 18 | 15 | 15 | 15
  ≥3-Fold, <4-Fold | 2 | 2 | 0 | 5 | 3 | 6 | 1 | 4 | 3 | 4
  ≥4-Fold | 1 | 1 | 2 | 1 | 2 | 2 | 8 | 7 | 8 | 3

42. Secondary Outcome: Fold Change in IgG Response to BCH0785 Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 36 | 35 | 35 | 36 | 42 | 31 | 27 | 26 | 20 | 32
  ≥2-Fold, <3-Fold | 9 | 11 | 8 | 6 | 4 | 7 | 8 | 14 | 17 | 11
  ≥3-Fold, <4-Fold | 1 | 0 | 0 | 4 | 2 | 5 | 6 | 2 | 1 | 1
  ≥4-Fold | 2 | 3 | 5 | 1 | 1 | 3 | 6 | 6 | 8 | 4

43. Secondary Outcome: Fold Change in IgG Response to StkP Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 38 | 35 | 42 | 38 | 41 | 22 | 21 | 22 | 24 | 35
  ≥2-Fold, <3-Fold | 6 | 9 | 4 | 7 | 6 | 16 | 15 | 18 | 14 | 9
  ≥3-Fold, <4-Fold | 2 | 0 | 0 | 2 | 2 | 3 | 4 | 0 | 4 | 2
  ≥4-Fold | 2 | 5 | 2 | 0 | 0 | 5 | 7 | 8 | 4 | 2

44. Secondary Outcome: Fold Change in IgG Response to PcpA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 37 | 42 | 40 | 39 | 33 | 30 | 32 | 35 | 26 | 23
  ≥2-Fold, <3-Fold | 7 | 3 | 4 | 5 | 10 | 9 | 7 | 7 | 9 | 15
  ≥3-Fold, <4-Fold | 1 | 3 | 0 | 1 | 0 | 2 | 3 | 3 | 3 | 1
  ≥4-Fold | 3 | 1 | 4 | 2 | 6 | 5 | 5 | 3 | 8 | 9

45. Secondary Outcome: Fold Change in IgG Response to SPWCA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 45 | 42 | 42 | 45 | 44 | 38 | 40 | 36 | 31 | 41
  ≥2-Fold, <3-Fold | 2 | 6 | 4 | 1 | 4 | 6 | 6 | 10 | 12 | 6
  ≥3-Fold, <4-Fold | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
  ≥4-Fold | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 1

46. Secondary Outcome: Fold Change in IgG Response to PiuA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 39 | 35 | 37 | 37 | 46 | 30 | 27 | 23 | 24 | 39
  ≥2-Fold, <3-Fold | 5 | 7 | 6 | 9 | 0 | 11 | 14 | 18 | 14 | 5
  ≥3-Fold, <4-Fold | 3 | 5 | 2 | 1 | 3 | 3 | 2 | 0 | 2 | 2
  ≥4-Fold | 1 | 2 | 3 | 0 | 0 | 2 | 4 | 7 | 6 | 2

47. Secondary Outcome: Fold Change in IgG Response to PiaA Pneumococcal Protein
Description: Measured using MSD
Time Frame: 28 days (post-vaccination 1) and 56 days (post-vaccination 2)
Measure: Count of Participants; unit: Participants
Arm/Group | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 1 | Active Control Only: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49 | 46 | 47 | 48 | 46 | 48
Participants
  <2-Fold | 39 | 36 | 39 | 35 | 41 | 25 | 25 | 22 | 24 | 32
  ≥2-Fold, <3-Fold | 7 | 8 | 6 | 8 | 4 | 12 | 12 | 18 | 13 | 8
  ≥3-Fold, <4-Fold | 0 | 3 | 2 | 2 | 2 | 4 | 4 | 2 | 4 | 3
  ≥4-Fold | 2 | 2 | 1 | 2 | 2 | 5 | 6 | 6 | 5 | 5

48. Secondary Outcome: Number/Percentage of Adult Subjects With Neutralizing Antibody Response to Pneumolysin
Description: Functional antibody responses to Ply (pneumolysin) were assessed using a toxin neutralization assay based on the ability of antibodies to neutralize wild-type Ply-induced lysis of rabbit red blood cells. Briefly, serial 2-fold dilutions (starting at 1/5 dilution) of human serum samples were added together with wild-type Ply in 96-well plates. Rabbit red blood cells were then added and following incubation supernatants removed and transferred to new 96-well plates and absorbance measured at 540 nm using a spectrophotometer plate reader. The mean A450 nm blank value was subtracted by 10% to obtain the Plate Specific Cut Point for each plate. Each sample was categorized as negative (<1/20) or positive (with titer between 1/20 and 1/320).
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Measure: Count of Participants; unit: Participants
Groups:
- PATH-wSP (600 mcg): Baseline: Subjects receiving 600 mcg PATH-wSP: levels pre-vaccination
- PATH-wSP (600 mcg): Vaccination 1: Subjects receiving 600 mcg PATH-wSP: levels after first vaccination
- PATH-wSP (600 mcg): Vaccination 2: Subjects receiving 600 mcg PATH-wSP: levels after second vaccination
- PATH-wSP (1000 mcg): Baseline: Subjects receiving 1000 mcg PATH-wSP: levels pre-vaccination
- PATH-wSP (1000 mcg): Vaccination 1: Subjects receiving 1000 mcg PATH-wSP: levels after first vaccination
- PATH-wSP (1000 mcg): Vaccination 2: Subjects receiving 1000 mcg PATH-wSP: levels after second vaccination
- Saline: Baseline: Subjects receiving saline placebo injection: levels pre-vaccination
- Saline: Vaccination 1: Subjects receiving saline placebo injection: levels after vaccination 1
- Saline: Vaccination 2: Subjects receiving saline placebo injection: levels after vaccination 2
Arm/Group | PATH-wSP (600 mcg): Baseline | PATH-wSP (600 mcg): Vaccination 1 | PATH-wSP (600 mcg): Vaccination 2 | PATH-wSP (1000 mcg): Baseline | PATH-wSP (1000 mcg): Vaccination 1 | PATH-wSP (1000 mcg): Vaccination 2 | Saline: Baseline | Saline: Vaccination 1 | Saline: Vaccination 2
Number analyzed (Participants) | 18 | 18 | 17 | 18 | 18 | 18 | 17 | 17 | 17
Participants
  <1:20 | 3 | 3 | 2 | 5 | 3 | 3 | 2 | 3 | 4
  1:20 | 7 | 4 | 2 | 7 | 8 | 3 | 10 | 7 | 6
  1:40 | 5 | 5 | 4 | 5 | 5 | 8 | 5 | 7 | 7
  1:80 | 3 | 5 | 6 | 1 | 2 | 4 | 0 | 0 | 0
  1:160 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Number/Percentage of Toddler Subjects With Neutralizing Antibody Response to Pneumolysin
Description: as for outcome 48
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Measure: Count of Participants; unit: Participants
Groups:
- PATH-wSP (300 mcg)+Active Control: Baseline: Subjects receiving 300 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: pre-vaccination
- PATH-wSP (300 mcg)+Active Control: Vaccination 1: Subjects receiving 300 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 1
- PATH-wSP (300 mcg)+Active Control: Vaccination 2: Subjects receiving 300 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 2
- PATH-wSP (300 mcg)+Saline: Baseline: Subjects receiving 300 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: pre-vaccination
- PATH-wSP (300 mcg)+Saline: Vaccination 1: Subjects receiving 300 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: after vaccination 1
- PATH-wSP (300 mcg)+Saline: Vaccination 2: Subjects receiving 300 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: after vaccination 2
- PATH-wSP (600 mcg)+Active Control: Baseline: Subjects receiving 600 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: pre-vaccination
- PATH-wSP (600 mcg)+Active Control: Vaccination 1: Subjects receiving 600 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 1
- PATH-wSP (600 mcg)+Active Control: Vaccination 2: Subjects receiving 600 mcg PATH-wSP in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 2
- PATH-wSP (600 mcg)+Saline: Baseline: Subjects receiving 600 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: pre-vaccination
- PATH-wSP (600 mcg)+Saline: Vaccination 1: Subjects receiving 600 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: after Vaccination 1
- PATH-wSP (600 mcg)+Saline: Vaccination 2: Subjects receiving 600 mcg PATH-wSP in the left thigh and two injections of saline placebo in the right thigh: after Vaccination 2
- Active Control Only: Baseline: Subjects receiving saline placebo injection in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: pre-vaccination
- Active Control Only: Vaccination 1: Subjects receiving saline placebo injection in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 1
- Active Control Only: Vaccination 2: Subjects receiving saline placebo injection in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh: after vaccination 2
Arm/Group | PATH-wSP (300 mcg)+Active Control: Baseline | PATH-wSP (300 mcg)+Active Control: Vaccination 1 | PATH-wSP (300 mcg)+Active Control: Vaccination 2 | PATH-wSP (300 mcg)+Saline: Baseline | PATH-wSP (300 mcg)+Saline: Vaccination 1 | PATH-wSP (300 mcg)+Saline: Vaccination 2 | PATH-wSP (600 mcg)+Active Control: Baseline | PATH-wSP (600 mcg)+Active Control: Vaccination 1 | PATH-wSP (600 mcg)+Active Control: Vaccination 2 | PATH-wSP (600 mcg)+Saline: Baseline | PATH-wSP (600 mcg)+Saline: Vaccination 1 | PATH-wSP (600 mcg)+Saline: Vaccination 2 | Active Control Only: Baseline | Active Control Only: Vaccination 1 | Active Control Only: Vaccination 2
Number analyzed (Participants) | 46 | 46 | 46 | 47 | 47 | 47 | 48 | 48 | 48 | 47 | 47 | 46 | 48 | 48 | 48
Participants
  <1:20 | 20 | 19 | 14 | 18 | 10 | 11 | 17 | 14 | 6 | 14 | 7 | 6 | 27 | 21 | 19
  1:20 | 11 | 9 | 10 | 15 | 15 | 10 | 13 | 13 | 11 | 12 | 12 | 6 | 10 | 13 | 17
  1:40 | 10 | 8 | 9 | 8 | 14 | 14 | 13 | 14 | 16 | 14 | 10 | 13 | 6 | 11 | 6
  1:80 | 2 | 8 | 8 | 5 | 5 | 7 | 3 | 5 | 10 | 6 | 11 | 13 | 4 | 3 | 5
  1:160 | 1 | 2 | 4 | 0 | 2 | 5 | 2 | 1 | 3 | 1 | 6 | 5 | 1 | 0 | 0
  1:320 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 3 | 0 | 0 | 1

50. Other Pre Specified Outcome: Geometric Mean Concentration (GMCs) of PNC-IgG Serotypes Among Toddler Subjects
Description: GMCs of these IgG proteins were measured to assess potential interference of PATH-wSP with 10-valent pneumococcal conjugate vaccine (Synflorix). GMCs of Cohort 1 were measured at a different time point than those in Cohort 2, so results are presented separately.
Time Frame: 12 weeks (Cohort 1) and 4 weeks (Cohort 2) post-vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/mL
Groups:
- Cohort 1: PATH-wSP 300 mcg+Active Control: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- Cohort 1: PATH-wSP 300 mcg+Saline: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
  PATH-wSP: Streptococcus pneumoniae Whole Cell Vaccine adsorbed to Alum
  Saline: 0.9% Sodium Chloride Injection, USP
- Cohort 1: Active Control Only: A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
- Cohort 2 PATH-wSP 600 mcg+Active Control: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- Cohort 2: PATH-wSP 600 mcg+Saline: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
  PATH-wSP: Streptococcus pneumoniae Whole Cell Vaccine adsorbed to Alum
  Saline: 0.9% Sodium Chloride Injection, USP
- Cohort 2: Active Control Only: A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
  Synflorix: 1 dose (0.5 mL) contains:
  1 μg of each of the following pneumococcal polysaccharide serotypes:
  1, 5, 6B, 7F, 9V, 14, and 23 F
  And 3 μg of the following pneumococcal polysaccharide serotypes:
  4, 18C and 19F.
  The serotypes are conjugated to either:
  protein D (derived from Non-Typeable Haemophilus influenzae) carrier protein, tetanus toxoid carrier protein or diphtheria toxoid carrier protein
  Pentavac: Each PFS contains 0.5 ml (single dose):
  Diphtheria Toxoid 20 Lf to 30 Lf Tetanus Toxoid 2.5 Lf to 10 Lf B. Pertussis 4 IU HBsAg (rDNA) 10 mcg Purified capsular HIB Polysaccharide (PRP) Conjugated to Tetanus Toxoid (carrier protein) 10 mcg Adsorbed on Aluminium Phosphate, AL+++ 1.25 mg Preservative: Thiomersal 0.005 %
  Dose:
Arm/Group | Cohort 1: PATH-wSP 300 mcg+Active Control | Cohort 1: PATH-wSP 300 mcg+Saline | Cohort 1: Active Control Only | Cohort 2 PATH-wSP 600 mcg+Active Control | Cohort 2: PATH-wSP 600 mcg+Saline | Cohort 2: Active Control Only
Number analyzed (Participants) | 46 | 47 | 48 | 47 | 23 | 25
ug/mL
  PnC-IgG-ELISA type 1: number analyzed (Participants) | 46 | 46 | 48 | 45 | 23 | 25
  PnC-IgG-ELISA type 1 | 0.87 [0.72 to 1.06] | 0.18 [0.14 to 0.21] | 3.09 [2.50 to 3.83] | 0.25 [0.21 to 0.30] | 0.83 [0.64 to 1.08] | 2.47 [1.81 to 3.38]
  PnC-IgG-ELISA type 4 | 1.22 [1.01 to 1.47] | 0.28 [0.22 to 0.34] | 3.41 [2.93 to 3.96] | 0.36 [0.29 to 0.46] | 1.15 [0.89 to 1.50] | 2.59 [2.08 to 3.22]
  PnC-IgG-ELISA type 5 | 0.38 [0.32 to 0.45] | 0.17 [0.14 to 0.20] | 0.77 [0.64 to 0.92] | 0.19 [0.16 to 0.23] | 0.44 [0.33 to 0.58] | 0.77 [0.65 to 0.90]
  PnC-IgG-ELISA type 6B: number analyzed (Participants) | 45 | 46 | 48 | 47 | 23 | 25
  PnC-IgG-ELISA type 6B | 1.60 [1.33 to 1.92] | 0.69 [0.54 to 0.88] | 4.28 [3.48 to 5.27] | 0.95 [0.76 to 1.18] | 2.19 [1.62 to 2.94] | 3.68 [2.68 to 5.06]
  PnC-IgG-ELISA type 7F | 1.79 [1.48 to 2.16] | 0.60 [0.50 to 0.72] | 4.32 [3.63 to 5.13] | 0.72 [0.59 to 0.89] | 1.36 [1.04 to 1.79] | 3.57 [2.97 to 4.28]
  PnC-IgG-ELISA type 9V | 0.77 [0.65 to 0.91] | 0.26 [0.20 to 0.33] | 2.03 [1.73 to 2.38] | 0.29 [0.24 to 0.35] | 0.71 [0.51 to 0.97] | 1.57 [1.25 to 1.97]
  PnC-IgG-ELISA type 14: number analyzed (Participants) | 46 | 47 | 48 | 46 | 23 | 25
  PnC-IgG-ELISA type 14 | 3.16 [2.54 to 3.92] | 0.63 [0.50 to 0.78] | 8.62 [7.02 to 10.57] | 1.02 [0.79 to 1.33] | 3.20 [2.36 to 4.34] | 7.40 [5.37 to 10.20]
  PnC-IgG-ELISA type 18C: number analyzed (Participants) | 46 | 47 | 48 | 46 | 23 | 25
  PnC-IgG-ELISA type 18C | 1.51 [1.25 to 1.82] | 0.28 [0.22 to 0.35] | 3.52 [3.00 to 4.13] | 0.33 [0.27 to 0.41] | 1.31 [1.00 to 1.71] | 3.05 [2.43 to 3.82]
  PnC-IgG-ELISA type 19F: number analyzed (Participants) | 46 | 47 | 48 | 45 | 23 | 25
  PnC-IgG-ELISA type 19F | 4.62 [3.78 to 5.63] | 1.48 [1.08 to 2.02] | 10.93 [8.92 to 13.38] | 1.50 [1.17 to 1.93] | 4.76 [3.33 to 6.80] | 7.59 [5.10 to 11.29]
  PnC-IgG-ELISA type 23F: number analyzed (Participants) | 41 | 46 | 38 | 45 | 22 | 24
  PnC-IgG-ELISA type 23F | 0.98 [0.77 to 1.25] | 0.27 [0.21 to 0.35] | 2.76 [2.22 to 3.44] | 0.28 [0.21 to 0.37] | 0.97 [0.70 to 1.34] | 3.50 [2.60 to 4.70]

51. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Diptheria Booster Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: IU/mL
Groups:
- PATH-wSP 300 mcg+Active Control: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
- PATH-wSP 300 mcg+Saline: A single injection of PATH-wSP 300 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 300 mcg in the left thigh 8 weeks later.
  PATH-wSP: Streptococcus pneumoniae Whole Cell Vaccine adsorbed to Alum
  Saline: 0.9% Sodium Chloride Injection, USP
- PATH-wSP 600 mcg+Active Control: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of each of the two active comparator vaccines (Synflorix and Pentavac) in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
- PATH-wSP 600 mcg+Saline: A single injection of PATH-wSP 600 mcg in the left thigh and a single injection of saline in the right thigh along with a separate single injection of saline in the right thigh. These 3 injections are followed by a single injection of PATH-wSP 600 mcg in the left thigh 8 weeks later.
  PATH-wSP: Streptococcus pneumoniae Whole Cell Vaccine adsorbed to Alum
  Saline: 0.9% Sodium Chloride Injection, USP
- Active Control Only: A single injection of saline in the left thigh and a single injection of each of the two active comparator vaccines in the right thigh. These 3 injections are followed by a single injection of saline in the left thigh 8 weeks later.
  Synflorix: 1 dose (0.5 mL) contains:
  1 μg of each of the following pneumococcal polysaccharide serotypes:
  1, 5, 6B, 7F, 9V, 14, and 23 F
  And 3 μg of the following pneumococcal polysaccharide serotypes:
  4, 18C and 19F.
  The serotypes are conjugated to either:
  protein D (derived from Non-Typeable Haemophilus influenzae) carrier protein, tetanus toxoid carrier protein or diphtheria toxoid carrier protein
  Pentavac: Each PFS contains 0.5 ml (single dose):
  Diphtheria Toxoid 20 Lf to 30 Lf Tetanus Toxoid 2.5 Lf to 10 Lf B. Pertussis 4 IU HBsAg (rDNA) 10 mcg Purified capsular HIB Polysaccharide (PRP) Conjugated to Tetanus Toxoid (carrier protein) 10 mcg Adsorbed on Aluminium Phosphate, AL+++ 1.25 mg Preservative: Thiomersal 0.005 %
  Dose:
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
IU/mL | 7.73 [6.38 to 9.36] | 0.25 [0.20 to 0.32] | 7.71 [6.48 to 9.19] | 0.27 [0.22 to 0.33] | 9.39 [7.90 to 11.15]

52. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Hepatitis B Booster Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: mIU/mL
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
mIU/mL | 784.78 [532.71 to 11156.12] | 149.86 [83.65 to 268.47] | 695.14 [546.72 to 883.84] | 135.79 [84.93 to 217.11] | 815.39 [705.76 to 942.04]

53. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Haemophilus Influenzae Type b (Hib) Booster Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/mL
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
ug/mL | 41.05 [29.61 to 56.92] | 1.68 [1.20 to 2.34] | 39.06 [30.70 to 49.68] | 1.23 [0.81 to 1.88] | 37.45 [25.82 to 54.32]

54. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Pertussis FHA and Pertussis Toxin Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: IU/mL
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
IU/mL
  Pertussis FHA | 85.12 [73.07 to 99.17] | 6.70 [5.48 to 8.21] | 68.23 [57.45 to 81.05] | 10.47 [8.40 to 13.05] | 90.65 [73.87 to 111.23]
  Pertussis Toxin | 145.11 [121.66 to 173.08] | 19.38 [15.13 to 24.81] | 131.23 [105.83 to 162.73] | 18.79 [13.55 to 26.07] | 124.39 [96.63 to 160.11]

55. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Pertussis Fimbriae Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: U/mL
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
U/mL | 753.63 [582.34 to 975.30] | 45.75 [32.98 to 63.47] | 460.73 [328.95 to 645.31] | 37.99 [27.75 to 52.00] | 503.25 [383.05 to 661.17]

56. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) Ratio of Tetanus Booster Immune Response Among Toddler Subjects
Description: GMCs of these proteins were measured to assess potential interference of PATH-wSP with Pentavac booster dose.
Time Frame: 12 weeks post vaccination 1
Population: The number analyzed may differ between proteins because of insufficient samples.
Measure: Geometric Mean (90% Confidence Interval); unit: IU/mL
Arm/Group | PATH-wSP 300 mcg+Active Control | PATH-wSP 300 mcg+Saline | PATH-wSP 600 mcg+Active Control | PATH-wSP 600 mcg+Saline | Active Control Only
Number analyzed (Participants) | 48 | 49 | 48 | 47 | 49
IU/mL | 21.83 [18.94 to 25.17] | 1.15 [0.93 to 1.43] | 21.64 [19.01 to 24.62] | 1.27 [1.03 to 1.55] | 21.92 [18.95 to 25.35]

ADVERSE EVENTS:
Time Frame: 4 weeks post-vaccination
Description: Subjects returned to the clinic 1 week post each vaccination and at 4 weeks after the final vaccination for assessment of solicited reactogenicity, targeted physical examination, vital signs, laboratory assessment, immunology testing, and evaluation for unsolicited AEs and concomitant medication use.
Arm/Group | Adult Cohort: PATH-wSP (600 mcg) | Adult Cohort: PATH-wSP (1000 mcg) | Adult Cohort: Saline | Toddler Cohort: PATH-wSP (300 mcg)+Active Control | Toddler Cohort: PATH-wSP (300 mcg)+Saline | Toddler Cohort: PATH-wSP (600 mcg)+Active Control | Toddler Cohort: PATH-wSP (600 mcg)+Saline | Toddler Cohort: Active Control Only
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 1/50 | 0/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 0/18 | 6/50 | 2/50 | 2/50 | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 18/18 | 16/18 | 17/18 | 50/50 | 47/50 | 48/50 | 48/50 | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Cohort: PATH-wSP (600 mcg) (N=18) | Adult Cohort: PATH-wSP (1000 mcg) (N=18) | Adult Cohort: Saline (N=18) | Toddler Cohort: PATH-wSP (300 mcg)+Active Control (N=50) | Toddler Cohort: PATH-wSP (300 mcg)+Saline (N=50) | Toddler Cohort: PATH-wSP (600 mcg)+Active Control (N=50) | Toddler Cohort: PATH-wSP (600 mcg)+Saline (N=50) | Toddler Cohort: Active Control Only (N=50)
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic intracranial hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Cohort: PATH-wSP (600 mcg) (N=18) | Adult Cohort: PATH-wSP (1000 mcg) (N=18) | Adult Cohort: Saline (N=18) | Toddler Cohort: PATH-wSP (300 mcg)+Active Control (N=50) | Toddler Cohort: PATH-wSP (300 mcg)+Saline (N=50) | Toddler Cohort: PATH-wSP (600 mcg)+Active Control (N=50) | Toddler Cohort: PATH-wSP (600 mcg)+Saline (N=50) | Toddler Cohort: Active Control Only (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 10 | 4 | 7 | 5 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1 | 0 | 1 | 2 | 2
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 3 | 5 | 6 | 3 | 8 | 9
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 3 | 1 | 1
Dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 3 | 0 | 0 | 5 | 8 | 18 | 10 | 8
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 15 | 13 | 6 | 8 | 16
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 2 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Hepatobiliary (General disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 2
Pyrexia (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 3 | 5 | 4 | 11
Injection site pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 3 | 1 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 12 | 6 | 10 | 6 | 10
Malaria (Infections and infestations) | 3 | 5 | 6 | 20 | 26 | 15 | 17 | 16
Septic rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen increased (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4 | 5 | 6 | 5 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 2 | 6 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 6 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 3 | 5 | 0 | 3 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 2 | 2 | 5 | 7 | 0 | 0 | 3
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 8 | 41 | 39 | 44 | 43 | 43
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 8 | 6 | 0
Body tinea (Infections and infestations) | 1 | 0 | 1 | 0 | 3 | 6 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 10 | 3 | 3 | 6 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 5 | 11 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 3 | 5 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No